CLINICAL TRIAL: NCT04451525
Title: REal-World Analyses of Stroke - Thrombus Occlusion REtrieval
Acronym: "RESTORE"
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL11012
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Acute Ischemic Stroke; Vessel Occlusion; Stroke; Ischemic
Keywords: Mechanical Thrombectomy, Aspiration, SOFIA®, Direct Aspiration, ERIC®
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Cohort I: Cohort I will focus on data collection on the SOFIA® Flow Plus 6F Aspiration Catheter used with the direct aspiration as first line treatment technique with the intent to evaluate per prespecified endpoints.
  Interventions: Device: MicroVention Mechanical Thrombectomy Devices as first-line treatment
- Cohort II: Cohort II will focus on data collection on MicroVention devices used for acute ischemic stroke treatment with the intent to evaluate standard outcomes while also generating additional research questions for analysis based on data collected.
  Interventions: Device: MicroVention Mechanical Thrombectomy Devices as first-line treatment

INTERVENTIONS:
Device: MicroVention Mechanical Thrombectomy Devices as first-line treatment — Patient will be treated with mechanical thrombectomy at the direction of the treating physician

SUMMARY:
To collect real-world evidence allowing assessment of functional, imaging, and safety outcomes of MicroVention market-released acute ischemic stroke devices when used at the direction of the treating physician.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single arm, observational, Real World Evidence (RWE) post-market study with two cohorts.

The primary objective of Cohort I of the RESTORE study is to determine the proportion of subjects achieving successful revascularization (mTICI ≥ 2b) with the SOFIA® Flow Plus 6F Aspiration Catheter when used in conjunction with the direct aspiration as first line treatment technique for patients with acute ischemic stroke in the anterior circulation based on collection of real-world evidence data. Secondary objectives include the evaluation of good functional outcome (defined as mRS ≤ 2 at day 90), revascularization time, and procedure related major neurological complications, all based on real-world evidence data collected.

The objective of Cohort II of the study is to evaluate standard outcomes such as successful revascularization (mTICI ≥ 2b), good functional outcome (defined as mRS ≤ 2 at day 90), revascularization time, and procedure related major neurological complications based on real-world evidence data. Additional outcomes may be defined and research questions generated based on review of the collected data.

ELIGIBILITY:
Cohort I:

Inclusion Criteria:

1. Patient is ≥ 21 and ≤ 85 years of age.
2. Patient has a pre-morbid mRS ≤ 1.
3. Neuroimaging (CT/CTA and/or MR/MRA collected at no more than 90 minutes prior to groin puncture) demonstrates large vessel proximal occlusion (distal ICA through MCA bifurcation).
4. Patient has an NIHSS score ≥ 5 at time of intervention.
5. Symptom onset is within 8 hours of when groin puncture can be achieved.
6. Patient will undergo treatment via femoral access and the decision to use femoral access has been made by the treating physician outside the context of the RESTORE study and prior to study enrollment.
7. Patient will be treated using the direct aspiration as first line treatment technique and the decision to use this technique and the study device has been made by the treating physician outside the context of the RESTORE study and prior to study enrollment.
8. Patient or patient's legally authorized representative (LAR) has provided written informed consent.
9. Patient is considered by the treating physician to be available for and able to complete all follow-up visits with a trained site investigator.

Exclusion Criteria:

1. Inability to obtain written informed consent.
2. Patient is < 21 or > 85 years of age.
3. Patient has a pre-morbid mRS ≥ 2.
4. More than 8 hours have passed since symptom onset.
5. Severe unilateral or bilateral carotid artery stenosis or dissection requiring stent treatment.
6. Presence of a pre-existing large territory infarction.
7. Absent femoral pulses or other condition preventing femoral access.
8. Patient has vascular anatomy/tortuosity or other vascular disease preventing access to the target occlusion or that will likely result in unstable access.
9. Patient is pregnant.
10. Known or suspected pre-existing/chronic large vessel occlusion in the symptomatic territory.
11. Patient has known, untreatable hypersensitivity to contrast dye, iodine or any component of the treatment device that cannot be medically controlled.
12. The intracranial occlusion is suspected to be chronic based on past imaging, clinical history, or clinical judgment.
13. Patient has a severe or life-threatening comorbidity that could confound study results, or that will render the procedure unlikely to benefit the patient.
14. Patient is unable to complete scheduled follow-up assessments due to comorbidities, geographical limitations, or a life expectancy of less than 3 months.
15. Patient is enrolled in another device or drug study in which participation could confound study results.
16. Imaging (CT or MR) exclusion criteria:

    * Presence of intracerebral hemorrhage as evidenced on initial imaging
    * Ischemic changes in the posterior circulation territories (including the vertebra-basilar and posterior cerebral arteries)
    * Significant mass effect with midline shift
    * Evidence of intracranial tumor
    * Baseline ischemic core lesion >50 cc
    * Involvement of > 1/3 of the middle cerebral artery territory
    * ASPECTS <6 (hemispheric sulcal effacement and/or loss of grey-white differentiation alone are not contraindications for treatment)

Cohort II:

Inclusion Criteria:

1. Neuroimaging (CT/CTA and/or MR/MRA) demonstrates intracranial vessel occlusion.
2. Symptom onset is within 24 hours of when arterial access puncture can be achieved.
3. Patient will be treated using an FDA-cleared/approved and market-released MicroVention mechanical thrombectomy device as the initial, primary treatment device and the decision to use this device has been made by the treating physician outside the context of the RESTORE study and prior to study enrollment.

   Note: For the purposes of this protocol, ancillary/accessory devices such as balloon guide catheters and other access devices are not considered primary treatment devices. Further, devices used for rescue following attempt of a different primary treatment device are not considered initial primary treatment devices.
4. Patient or patient's legally authorized representative (LAR) has provided written informed consent within 48 hours of procedure.

Exclusion Criteria:

1. Inability to obtain written informed consent within 48 hours of procedure.
2. Patient is enrolled in another device or drug study in which participation could confound study results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with acute ischemic stroke in the cerebral circulation who will be treated with mechanical thrombectomy at the direction of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 710 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Cohort I: Proportion of subjects achieving mTICI ≥ 2b revascularization based on independent core lab assessment | During the procedure

SECONDARY OUTCOMES:
Proportion of subjects with good functional outcome defined as mRS ≤ 2 | 90 days
Occurrence of procedure related serious adverse events | During the procedure through study completion at 90 days
Occurrence of sICH within 24 hours | 24 hours post-operative
Occurrence of embolization to new territories (ENT) | During the procedure
Presence of vasospasm involving the accessed vascular tree | During the procedure through 24 hours post-operative
Mortality at day 90 | 90 days post-procedure
Proportion of subjects achieving mTICI ≥ 2b revascularization after first line aspiration treatment | During the procedure
Number of passes to achieve mTICI ≥ 2b revascularization with first line aspiration treatment | During the procedure
Proportion of subjects achieving mTICI ≥ 2b revascularization after first aspiration pass | During the procedure
Time from groin puncture to initial contact of clot with aspiration catheter | During the procedure
Time from groin puncture to achieve mTICI ≥ 2b using first line aspiration treatment | During the procedure
Technical success using the MicroVention BOBBY Balloon Guide Catheter based on successful placement at the target location and successful balloon inflation | During the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Gandhi, MBBS, MD, Principal Investigator — University of Maryland, Baltimore; Syed Zaidi, MD, Principal Investigator — ProMedica Toledo
Locations (37):
- United States (37):
  - Pacific Neuroscience Institute (Providence), Burbank, California
  - Mercy San Juan - Dignity Health Research Institute, Carmichael, California
  - Kaiser Permanente, Northern California, Redwood City, California
  - UCHealth Memorial, Colorado Springs, Colorado
  - Memorial Healthcare System, Hollywood, Florida
  - Tampa General Hospital, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Javon Bea Hospital, Rockford, Illinois
  - Goodman Campbell Brain and Spine, Carmel, Indiana
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Ascension Borgess, Kalamazoo, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health West, Wyoming, Michigan
  - Allina Health (Abbott Northwestern Hospital), Minneapolis, Minnesota
  - SSM Health, Bridgeton, Missouri
  - University of Missouri, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - HMH Jersey Shore University Medical Center, Neptune City, New Jersey
  - Northshore University Hospital - Northwell, Manhasset, New York
  - Mt. Sinai Health System, New York, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Montefiore, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - ProMedica Toledo, Toledo, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Geisinger, Danville, Pennsylvania
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
  - Prisma Health Upstate, Greenville, South Carolina
  - Sanford Medical Center, Sioux Falls, South Dakota
  - Semmes Murphy Clinic, Memphis, Tennessee
  - INOVA, Falls Church, Virginia
  - Swedish Health Services, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided